CLINICAL TRIAL: NCT03165578
Title: Neural Correlates of Neurofeedback Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frank Scharnowski (Other)
Responsible Party: Sponsor-Investigator, Frank Scharnowski, Prof. Dr., Psychiatric University Hospital, Zurich
Organization: Psychiatric University Hospital, Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PsychiatricUHZ
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Nicotine Dependence; Depression; PTSD
MeSH Terms: conditions — Tobacco Use Disorder; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback (Experimental): Neurofeedback training.
  Interventions: Other: Neurofeedback training
- Sham Feedback (Sham Comparator): Sham controlled neurofeedback training. Subjects in the sham control group will undergo the same procedure as subjects in the experimental group, but instead of being shown feedback derived from their own brain activity, they will be shown replayed feedback values from a randomly chosen subject of the experimental group.
  Interventions: Other: Sham Feedback

INTERVENTIONS:
Other: Neurofeedback training — In a neurofeedback setting, brain activity is measured non-invasively, the brain imaging data is analyzed in real-time, and then feedback regarding the current level of brain activity is provided to the subject.
  Arms: Neurofeedback
Other: Sham Feedback — Sham controlled neurofeedback training. Subjects in the sham control group will undergo the same procedure as subjects in the experimental group, but instead of being shown feedback derived from their own brain activity, they will be shown replayed feedback values from a randomly chosen subject of the experimental group.
  Arms: Sham Feedback

SUMMARY:
The objective of the present study is to identify brain networks in patients that contribute to successfully learning self-regulation with real-time fMRI.

DETAILED DESCRIPTION:
Neurofeedback has been established as a promising non-pharmacological therapeutic approach. However, patients differ in their ability to learn control over their own brain activity with neurofeedback. It is thus crucial to understand the brain networks that mediate learned self-regulation with real-time fMRI. The objective of the present study is thus to identify brain networks in patients that contribute to successfully learning self-regulation with real-time fMRI. To achieve this goal, patients suffering from depression, post-traumatic stress disorder, and nicotine addiction will be trained to improve their self-regulation skills using established real-time fMRI neurofeedback protocols.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic resonance imaging compatibility.
* DSM-V diagnosis of major depressive disorder, post-traumatic stress disorder, or nicotine addiction, respectively.

Exclusion Criteria:

* Other physical or psychiatric disorders.
* Current substance abuse.
* Exclusion criteria applicable to MRI (metallic implants, claustrophobia, epilepsy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
brain patterns that mediate learning self-regulation in patients with fMRI neurofeedback | 12 months
  Functional MRI data will be analysed using a whole brain mixed effect analysis across all subjects that compares brain patterns during self-regulation and baseline.

SECONDARY OUTCOMES:
neurofeedback learning success | 12 months
  Increased self-regulation skills will be assessed by a comparison of the slopes of the neurofeedback learning curves between subjects in the experimental group vs. the sham control group.
behavioral consequences of neurofeedback training | 12 months
  Behavioral outcome measures (questionnaires, standard clinical assessments) will be compared between subjects in the experimental group vs. the sham control group.
maintenance of learned self-regulation | 12 months
  An assessment of learned self-regulation (i.e. increase of the feedback signal in up-regulation compared to baseline blocks) in follow-up scanning sessions that will take place 6 months and 1 year after neurofeedback training. This will be a measure of how well learned self-regulation can be maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scharnowski, Prof. Dr., Principal Investigator — Hospital of Psychiatry, University of Zurich
Locations (1):
- Hospital of Psychiatry, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No